CLINICAL TRIAL: NCT05443503
Title: Stanford Spine Keeper (Who Has Your Back) - A Lifestyle Modification Program for Management of Chronic Low Back Pain
Brief Title: Stanford Spine Keeper - Managing Your Low Back Pain
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Software re-development in progress
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Matthew W Smuck, Assistant Professor, Orthopaedic Surgery Director, Stanford Interventional Spine Center Director, PM&R Spine Fellowship, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 43204
Record Dates: First submitted 2018-12-04; First posted 2022-07-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Patients can choose among or choose to be assigned to 2 tracks for management for their low back pain. The tracks include one focused on relaxation and symptom management, and another track on increasing activity. Each include educational material adapted from various sources from North America Spine Society (NASS), Center for Disease Control (CDC), National Institue of Health (NIH).
  Patients will stay in track for 28 days. After this, they may choose to remain in track and continue to perform maintenance activities or to engage in a different track.
  Interventions: Other: Mobile health applications (mHealth apps) based intervention

INTERVENTIONS:
Other: Mobile health applications (mHealth apps) based intervention — Patients can choose among or choose to be assigned to 2 tracks for management for their low back pain. The tracks include one focused on relaxation and symptom management, and another track on increasing activity. Each include educational material adapted from various sources from North America Spine Society (NASS), Center for Disease Control (CDC), National Institue of Health (NIH). Patients will stay in track for 28 days. After this, they may choose to remain in track and continue to perform maintenance activities or to engage in a different track.
  Other Names: Stanford SpineKeeper

SUMMARY:
Mobile health applications (mHealth apps) are transforming medical research and intervention by allowing constant, instantaneous and personalized access to patients. The investigators have designed a mHealth app (Stanford SpineKeeper) utilizing the Apple ResearchKit and HealthKit platform, which is an open source software framework designed Apple Inc to be used by medical researchers to use for research purposes. The investigators will assess whether a multidisciplinary intervention delivered through the application can help improve quality of life and minimize symptoms in patients with chronic low back pain.

DETAILED DESCRIPTION:
The purpose of this study is to assess whether a mHealth app based intervention can improve symptoms and quality of life in human subjects. Access to human subjects is critical to the success of this project.

Recruitment:

Participants will be recruited via the Apple ResearchKit platform. Interested participants who answers "yes" to the questions "Are you having low back pain?" and "Have your back pain been an ongoing problem for 6 months or longer?" are eligible to download the mobile phone application and participate. Patients will provide electronic informed consent via the mobile application . A phone number will be provided for potential participants to call to speak to a live representative.

Materials

App Design:

The investigators designed the mobile phone application to be compatible with the Apple Inc (iPhone operating system [iOS] 8 or 9) platform - ResearchKit. Our app was based on codes from another Stanford approved ResearchKit study - MyHeart Counts. The ResearchKit platform is set up to help researchers design applications capable of performing HIPAA compliant informed consent, surveys, active tasks, account creation, and passcode pin entry. As in the original MyHeart Counts app, the smartphone consent process used here have been adapted from an opensource toolkit developed by Sage Bionetworks in collaboration with the Electronic Data Methods forum of the AHRQ (Agency for Healthcare Research & Quality). The consent process have previously been reviewed with faculty in the Stanford Center for Biomedical Ethics.

Intervention:

Patients can choose among or choose to be assigned to 2 tracks for management for their low back pain. The tracks include one focused on relaxation and symptom management, and another track on increasing activity. Each include educational material adapted from various sources from North America Spine Society (NASS), Center for Disease Control (CDC), National Institue of Health (NIH).

Patients will stay in track for 28 days. After this, they may choose to remain in track and continue to perform maintenance activities or to engage in a different track.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported "yes" to the question "Have you ever had low back pain for 6 months?"
2. Ownership of an iPhone with an updated operating system (iOS 8 or 9) compatible with Apple ResearchKit with internet connectivity.
3. Self-reported aged 18 years and older with medical-decision making capacity.
4. Literacy in the English language

Exclusion Criteria:

1. Any serious chronic medical issues (severe cardiac or pulmonary medical problems, cancer) that may limit ability to participate in physical therapy and home exercise.
2. Individuals who are pregnant, incarcerated, decisionally impaired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500000 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in reported functional marker profile | Recorded daily for 7 days starting at enrollment and after the completion of each 28-day cycle
  Qualitative assessment of back pain and quality of life using the Stanford Spine Keeper app, which utilizes the Recommended Minimum Dataset from NIH Task Force on Research Standards for Chronic Low Back.
Change in pain score | Recorded daily for 7 days starting at enrollment and after the completion of each 28-day cycle
  Patient-report pain rated on a 0-10 scale (0 = no pain, 10 = worst pain) using the Stanford Spine Keeper app, which utilizes the Recommended Minimum Dataset from NIH Task Force on Research Standards for Chronic Low Back.
Change in daily steps | Recorded daily for 7 days starting at enrollment and after the completion of each 28-day cycle
  Change in daily steps recorded using the Stanford Spine Keeper app, which utilizes the Recommended Minimum Dataset from NIH Task Force on Research Standards for Chronic Low Back.
Change in back range of motion | Recorded daily for 7 days starting at enrollment and after the completion of each 28-day cycle
  Change in back range of motion recorded using the Stanford Spine Keeper app, which utilizes the Recommended Minimum Dataset from NIH Task Force on Research Standards for Chronic Low Back.
Change in six-minute walk test | Recorded daily for 7 days starting at enrollment and after the completion of each 28-day cycle
  Change in six-minute walk test recorded using the Stanford Spine Keeper app, which utilizes the Recommended Minimum Dataset from NIH Task Force on Research Standards for Chronic Low Back.
Free-living physical activity log | Recorded daily for 7 days starting at enrollment and after the completion of each 28-day cycle
  Log of free-living (outside of the laboratory) physical activity recorded using the Stanford Spine Keeper app, which utilizes the Recommended Minimum Dataset from NIH Task Force on Research Standards for Chronic Low Back.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No